CLINICAL TRIAL: NCT02555397
Title: Phase 1 Trial of Oncolytic Adenovirus-Mediated Cytotoxic and Interleukin 12 Gene Therapy for Locally Recurrent Prostate Cancer After Definitive Radiotherapy
Brief Title: Phase 1 Trial of Interleukin 12 Gene Therapy for Locally Recurrent Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Farzan Siddiqui, Senior Staff Physician, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prostate Cancer (9829)
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Locally Recurrent; Gene Therapy; IL-12; Adenovirus
MeSH Terms: conditions — Prostatic Neoplasms; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single (Experimental): Single intraprostatic injection of Ad5-yCD/mutTKSR39rep-hIL12 adenovirus at a dose of 1 x 10e10 to 1 x 10e12 viral particles.
  Interventions: Biological: Ad5-yCD/mutTKSR39rep-hIL12

INTERVENTIONS:
Biological: Ad5-yCD/mutTKSR39rep-hIL12 — Single intraprostatic injection of Ad5-yCD/mutTKSR39rep-hIL12 on day 1

SUMMARY:
The primary purpose of this phase 1 study is to determine the dose-dependent toxicity and maximum tolerated dose (MTD) of oncolytic adenovirus-mediated cytotoxic and IL-12 gene therapy in men with locally recurrent prostate cancer after definitive radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven local recurrence of prostate cancer at least one year after the completion of definitive radiation therapy
* Evidence of biologically active disease as demonstrated by an unequivocally rising serum PSA level that is ≥ 2 ng/mL above the nadir
* PSA < 100 ng/mL
* Age ≥ 18 years
* Karnofsky performance status ≥ 70
* Negative lymph nodes as established by imaging (pelvic CT or pelvic MRI)
* No evidence of metastatic disease, as evaluated by bone scan and CT scan of the abdomen and pelvis.
* Subjects must have adequate baseline organ function as assessed by the the following laboratory values:
* Adequate renal function with serum creatinine ≤ 1.5 mg/dL
* Platelet count > 100,000/µL
* Absolute neutrophil count > 1,000/µL
* Hemoglobin > 10.0 g/dL
* Bilirubin > 1.5 mg/dL
* AST/SGOT and ALT/SGPT < 3.0 times upper limit of normal (ULN)
* Men of child-producing potential must be willing to consent to use effective contraception for at least 3 months after the gene therapy
* Subjects must possess the ability to give informed consent and express a willingness to meet all of the expected requirements of the protocol for the duration of the study

Exclusion Criteria:

* PSA ≥ 100 ng/mL
* Prostate volume > 100 cc
* Pathologically positive lymph nodes or nodes > 1.0 cm on imaging (nodes > 1.0 cm but biopsy negative are allowed.
* Evidence of M1 metastatic disease
* Prior invasive malignancy except for non-melanoma skin cancer within 5 years of enrollment. Subjects must be disease-free for > 5 years
* Prior radical prostatectomy, cryosurgery for prostate cancer, or bilateral orchiectomy for any reason
* If the subject had prior androgen deprivation therapy (ADT), the subject exhibited biochemical failure while on ADT
* Prior systemic chemotherapy for the study cancer (prior chemotherapy for a different cancer is allowed; however, subjects must be > 2 years post-completion of chemotherapy at the time of registration. Subjects on Proscar therapy must stop to be eligible)
* Major surgery planned within 3 months of registration
* Severe, active co-morbidity defined as:
* New York Health Association Class II or greater congestive heart failure or active ventricular arrhythmia requiring medication
* Chronic obstructive pulmonary disease (COPD) exacerbation or other respiratory illness requiring hospitalization within last 3 months or precluding study therapy at the time of registration
* Acute infection
* Previous history of liver disease including hepatitis
* Immunosuppressive therapy including systemic corticosteroids (use of inhaled and topical corticosteroids is permitted)
* Impaired immunity or susceptibility to serious viral infections
* Allergy to any product used in the protocol. If the subject has an allergy to Ciproflaxin, another antibiotic can be substituted at the discretion of the treating physician
* Serious medical or psychiatric illness or concomitant medication, which, in the judgement of the principal investigator, might interfere with the subject's ability to respond to or tolerate the treatment or complete the trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2024-01-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Background] Freytag SO, Barton KN, Zhang Y. Efficacy of oncolytic adenovirus expressing suicide genes and interleukin-12 in preclinical model of prostate cancer. Gene Ther. 2013 Dec;20(12):1131-9. doi: 10.1038/gt.2013.40. Epub 2013 Jul 11. PMID 23842593
- [Derived] Nyati S, Stricker H, Barton KN, Li P, Elshaikh M, Ali H, Brown SL, Hwang C, Peabody J, Freytag SO, Movsas B, Siddiqui F. A phase I clinical trial of oncolytic adenovirus mediated suicide and interleukin-12 gene therapy in patients with recurrent localized prostate adenocarcinoma. PLoS One. 2023 Sep 15;18(9):e0291315. doi: 10.1371/journal.pone.0291315. eCollection 2023. PMID 37713401

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral from the department of Radiation Oncology and the department of Urology at the Henry Ford Cancer Institute, Henry Ford Health System
Groups:
- AdV Dose: 1X10e10 vp: Single intraprostatic injection of Ad5-yCD/mutTKSR39rep-hIL12 adenovirus at a dose of 1 x 10e10 viral particles.
- AdV Dose: 3x10e10 vp: Single intraprostatic injection of Ad5-yCD/mutTKSR39rep-hIL12 adenovirus at a dose of 3 x 10e10 viral particles.
- AdV Dose: 1x10e11 vp: Single intraprostatic injection of Ad5-yCD/mutTKSR39rep-hIL12 adenovirus at a dose of 1x10e11 viral particles.
- AdV Dose: 3x10e11 vp: Single intraprostatic injection of Ad5-yCD/mutTKSR39rep-hIL12 adenovirus at a dose of 3x10e11 viral particles.
- AdV Dose: 1x10e12 vp: Single intraprostatic injection of Ad5-yCD/mutTKSR39rep-hIL12 adenovirus at a dose of 1x10e12 viral particles.
Period: Overall Study
Arm/Group | AdV Dose: 1X10e10 vp | AdV Dose: 3x10e10 vp | AdV Dose: 1x10e11 vp | AdV Dose: 3x10e11 vp | AdV Dose: 1x10e12 vp
Started | 3 | 3 | 3 | 3 | 3
Completed | 2 | 3 | 3 | 3 | 3
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AdV Dose: 1X10e10 vp | AdV Dose: 3x10e10 vp | AdV Dose: 1x10e11 vp | AdV Dose: 3x10e11 vp | AdV Dose: 1x10e12 vp | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 3 | 3 | 3 | 3 | 3 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 3 | 3 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 3 | 2 | 9
  White | 3 | 1 | 0 | 0 | 1 | 5
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Tumor Stage [Count of Participants; unit: Participants] — The stage of a cancer describes the size of a tumor and how far it has spread from where it originated. This is determined radiographically and pathologically. Higher staged cancer have a worse prognosis.
  Participants
    T1c | 3 | 2 | 2 | 1 | 3 | 11
    T2 | 0 | 1 | 1 | 1 | 0 | 3
    Not Detected | 0 | 0 | 0 | 1 | 0 | 1
Gleason Score [Number; unit: participants] — This grade is based on how abnormal the cells appear, with higher scores reflecting more abnormal cells.
  participants
    6 | 0 | 0 | 0 | 0 | 1 | 1
    7 | 0 | 2 | 1 | 0 | 1 | 4
    8 | 2 | 0 | 2 | 0 | 0 | 4
    9 | 0 | 1 | 0 | 2 | 0 | 3
    10 | 1 | 0 | 0 | 0 | 0 | 1
    Not assessed | 0 | 0 | 0 | 1 | 1 | 2
Pre-T PSA (ng/ml) [Count of Participants; unit: Participants]
  <4 ng/mL | 2 | 2 | 1 | 1 | 0 | 6
  >=4 and <10 ng/mL | 0 | 0 | 1 | 1 | 2 | 4
  >=10 ng/mL | 1 | 1 | 1 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Dose-dependent Toxicity
Time Frame: 30 days from date of adenovirus injection (defined as day 1)
Population: Arm specific adverse events
Measure: Number; unit: participants
Arm/Group | AdV Dose: 1X10e10 vp | AdV Dose: 3x10e10 vp | AdV Dose: 1x10e11 vp | AdV Dose: 3x10e11 vp | AdV Dose: 1x10e12 vp
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
participants
  Chills | 0 | 2 | 0 | 2 | 3
  Cytokine release syndrome | 0 | 0 | 0 | 0 | 0
  Mental status change | 0 | 0 | 0 | 0 | 1
  Dehydration | 0 | 0 | 0 | 0 | 2
  Diarrhea | 0 | 1 | 0 | 0 | 3
  Dyspnea | 1 | 0 | 0 | 1 | 0
  Fatigue | 2 | 1 | 0 | 1 | 3
  Fever | 0 | 0 | 0 | 2 | 3
  Flu-like symptoms | 0 | 1 | 0 | 1 | 1
  Hypotension | 0 | 0 | 0 | 0 | 0
  Nausea | 1 | 0 | 0 | 1 | 2
  Urinary frequency | 1 | 1 | 0 | 0 | 1
  Urinary incontinence | 0 | 0 | 0 | 0 | 0
  Urinary retention | 0 | 0 | 0 | 0 | 0
  Urinary tract pain | 0 | 0 | 0 | 0 | 0
  Vomiting | 1 | 0 | 0 | 1 | 0
  Malaise | 0 | 0 | 0 | 1 | 3
  Pain (thigh, kidney, head, fingers) | 0 | 0 | 0 | 1 | 3
  Anemia | 1 | 0 | 1 | 0 | 1
  Leukopenia | 0 | 2 | 2 | 1 | 3
  Lymphopenia | 3 | 1 | 2 | 2 | 3
  Neutropenia | 0 | 0 | 1 | 1 | 1
  Thrombocytopenia | 0 | 0 | 1 | 2 | 2
  ALT/SGPT increased | 1 | 1 | 1 | 1 | 1
  AST/SGOT increased | 0 | 0 | 1 | 1 | 2
  ALKP increased | 1 | 0 | 0 | 0 | 0
  CPK increased | 1 | 1 | 2 | 3 | 1
  Creatinine increased | 0 | 0 | 0 | 0 | 1
  GGT increased | 0 | 0 | 0 | 0 | 0
  Hypercalcemia | 1 | 0 | 1 | 1 | 0
  Hyperglycemia | 1 | 0 | 1 | 0 | 2
  Hypomagnesemia | 0 | 1 | 0 | 0 | 0
  Hyponatremia | 1 | 0 | 1 | 1 | 2

2. Secondary Outcome: PSA Response
Time Frame: 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Freedom From Biochemical/Clinical Failure (FFF)
Time Frame: 2 years
Reporting Status: Not Posted

4. Secondary Outcome: PSA Doubling Time (PSADT)
Time Frame: 2 years
Reporting Status: Not Posted

5. Secondary Outcome: Disease-specific and Overall Survival
Time Frame: 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Quality of Life (QOL)
Time Frame: 2 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Association Between the Primary and Secondary Outcomes and Immunological Endpoints Including Serum IL-12 and IFN-y Levels and NK Cell Cytolytic Activity
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All adverse events were collected through the primary toxicity endpoint (day 30)
Arm/Group | AdV Dose: 1X10e10 vp | AdV Dose: 3x10e10 vp | AdV Dose: 1x10e11 vp | AdV Dose: 3x10e11 vp | AdV Dose: 1x10e12 vp
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 2/3 | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AdV Dose: 1X10e10 vp (N=3) | AdV Dose: 3x10e10 vp (N=3) | AdV Dose: 1x10e11 vp (N=3) | AdV Dose: 3x10e11 vp (N=3) | AdV Dose: 1x10e12 vp (N=3)
Dyspnea (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 | 0 (0) | 1 (1) | 3 (3)
Urinary Frequency (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Diarrhea (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Chills (General disorders) | 0 (0) | 2 | 0 (0) | 2 | 3 (3)
Flu-Like Symptoms (General disorders) | 0 (0) | 1 | 0 (0) | 1 (1) | 1 (2)
Dehydration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 | 3
Nausea (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 | 2
Cytokine release syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental Status Change (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1
Hypotension (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (3) | 3 (6)
Lymphopenia (Blood and lymphatic system disorders) | 3 (5) | 1 (2) | 2 (3) | 2 (3) | 3 (7)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 2 (4)
ALT/SGPT increased (Blood and lymphatic system disorders) | 1 (6) | 1 (2) | 1 (1) | 1 (4) | 1 (2)
AST/SGOT increased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 2 (3)
ALKP increased (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Blood and lymphatic system disorders) | 1 (6) | 1 (1) | 2 (10) | 3 (4) | 1 (2)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 2 (7)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyponatremia (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 1 (1) | 1 (2) | 2 (6)
Hypomagnesemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (thigh, kidney, head, fingers) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Creatinine increase (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
GGT Increase (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT02555397/Prot_SAP_000.pdf